CLINICAL TRIAL: NCT04857619
Title: A Multicountry, Multicentre, Non-interventional, Retrospective Study to Describe the Real-world Treatment Patterns and Associated Outcomes in Patients With HER2-positive Unresectable or Metastatic Breast Cancer
Brief Title: Study to Describe the Real-world Treatment Patterns and Associated Outcomes in Patients With HER2-positive Unresectable or Metastatic Breast Cancer
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Other Study IDs: D9673R00005
Record Dates: First submitted 2021-04-21; First posted 2021-04-23 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Metastatic Breast Cancer
Keywords: Human epidermal growth factor receptor 2 - positive; Retrospective
MeSH Terms: conditions — Breast Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Retrospective: Patients who are diagnosed with HER2-positive unresectable or mBC and have received at least 1 LOT in the advanced setting will be included. Approximately a total of 570-830 patients will be enrolled in the study.
  Interventions: Other: None (Observational study)

INTERVENTIONS:
Other: None (Observational study) — The data on different types of treatment received by the patients, socio-demographics, and clinico-pathological characteristics and healthcare resource utilisation will be extracted from patients' medical records (both alive and deceased).
  Other Names: Observational study

SUMMARY:
This multicountry, multicenter, retrospective, non-interventional study involving patients diagnosed with HER2-positive unresectable or metastatic breast cancer mBC will be conducted to understand the demographic and clinico-pathological profile of the patients, diagnostic practices for human epidermal growth factor receptor 2 (HER2) status, current treatment landscape and sequencing of therapies, associated burden of toxicities with all lines of treatment (LOTs), and survival outcomes in the real-world setting.

DETAILED DESCRIPTION:
The study will involve patients diagnosed with HER2-positive unresectable or mBC since the earlier date between the date of trastuzumab emtansine ([T-DM1] Kadcyla) becoming available through reimbursement or patient access programme as a valid local treatment option or 01 January 2017 and who received at least 1 LOT. The data will be collected from the date of diagnosis of unresectable or mBC (index date) to the end of follow-up (ie, until death, the last medical record entry, or date of data extraction, whichever is earlier). The study will not have any study-specific patient visits or a longitudinal follow-up. All available data will be extracted from patients' medical records or obtained from patients themselves after obtaining an informed consent unless a waiver is granted by the local Institutional Review Board (IRB)/Institutional Ethics Committee (IEC)/Ethics Committee (EC). The informed consent may be obtained at the time of patients routine clinical care visit to the oncology centre. The data on different types of treatment received by the patients, socio-demographics, and clinico-pathological characteristics will be extracted from patients medical records up to the date informed consent was obtained.

This study will be conducted in non-US and non-European countries including Australia, Brazil, Hong Kong, Korea, Singapore and Taiwan. The total number of patients in the study will be approximately a minimum of 570 and a maximum of 830 patients. The study will be implemented at approximately 50 to 100 oncology centres spanning across 6 countries in the AstraZeneca (AZ) International Region (ie, non-US, non-European countries).

ELIGIBILITY:
Inclusion Criteria:

* Adult female or male patients ≥18 years old or 'adults' according to the age of majority as defined by the local regulations
* Patient or next of kin/legal representative willing and able to provide written informed consent according to the local regulations unless a waiver is granted by the local IRB/IEC/EC
* Patients' medical records showing a diagnosis of HER2-positive unresectable or mBC (can be either de novo advanced disease, progression or recurrence of previous early-stage HER2-positive BC) since the available date of T-DM1 (Kadcyla) through reimbursement or patient access programme as a valid local treatment option or 01 January 2017, whichever is earlier and with the availability of at least 12 months of follow-up data (from the date of diagnosis of unresectable or mBC) in the medical records at the participating site, unless patient died within the first 12 months of diagnosis
* Patients completing at least 1 LOT for HER2-positive unresectable or mBC

Exclusion Criteria:

* Patients with HER2-negative unresectable or mBC at index diagnosis
* Patients with a change in HER2 status from positive to negative at the progression from early-stage to advanced-stage disease (ie, shown on a repeat biopsy at diagnosis of advanced-stage disease) will be excluded (patients who change from HER2-positive to negative on repeat biopsy during treatment for advanced-stage disease may be included)
* Patients with concomitant cancer at the time of diagnosis of HER2-positive unresectable or mBC except for the non-metastatic non-melanoma skin cancers, or in situ, or benign neoplasms; a cancer is considered concomitant if it occurs within 5 years of HER2-positive breast cancer diagnosis
* Patients who at the time of data collection for this study are participating or have participated in an interventional study that remains blinded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will include patients who are diagnosed with HER2-positive unresectable or mBC and have received at least 1 LOT in the advanced setting.
Sampling Method: Non-Probability Sample
Enrollment: 763 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Percentage of patients receiving each treatment regimen with or without hormonal therapy in each LOT | Retrospective: from date of first diagnosis of unresectable or mBC (01 January 2017) to the end of follow-up (i.e., until death, the last medical record entry, or date of data extraction, whichever is the earliest) [Approximately 12 Months]
  Assessment of treatment patterns in patients diagnosed with HER2-positive unresectable or mBC. Line of treatment (LOT) is defined as one regimen, possibly a combination of several drugs, given from either the index diagnosis or disease progression until the treatment fails to control the disease, is not tolerated by the patient, the disease relapses/progresses, or death occurs.
Duration of therapy (DoT) for each regimen in each LOT | Retrospective: from date of first diagnosis of unresectable or mBC (01 January 2017) to the end of follow-up (i.e., until death, the last medical record entry, or date of data extraction, whichever is the earliest) [Approximately 12 Months]
  Assessment of length of time from initiation of therapy to permanent discontinuation. The DoT will be calculated as the time from the date of initiation of LOT to the stop of the treatment regimen for every LOT as per dates available in the medical record.
Percentage of patients receiving local and regional treatment for metastasis | Retrospective: from date of first diagnosis of unresectable or mBC (01 January 2017) to the end of follow-up (i.e., until death, the last medical record entry, or date of data extraction, whichever is the earliest) [Approximately 12 Months]
  Assessment of local and regional treatment for metastasis (radiotherapy and/or surgery), and bone protection therapy

SECONDARY OUTCOMES:
Demographic and clinico-pathological characteristics of patients with HER2-positive unresectable or mBC | Retrospective: from date of first diagnosis of unresectable or mBC (01 January 2017) to the end of follow-up (i.e., until death, the last medical record entry, or date of data extraction, whichever is the earliest) [Approximately 12 Months]
  Descriptive statistics will be used to describe socio-demographic and clinico-pathological characteristics for the overall study.
Real-world disease progression | Retrospective: from date of first diagnosis of unresectable or mBC (01 January 2017) to the end of follow-up (i.e., until death, the last medical record entry, or date of data extraction, whichever is the earliest) [Approximately 12 Months]
  Real-world disease progression of unresectable or mBC is defined as that documented in either the radiology report, pathology reports or clinician note as cancer progression.
Real-world progression free survival (rwPFS) | Retrospective: from date of first diagnosis of unresectable or mBC (01 January 2017) to the end of follow-up (i.e., until death, the last medical record entry, or date of data extraction, whichever is the earliest) [Approximately 12 Months]
  Real-world PFS is defined as the time from date of initiation of LOT to documented disease progression or death, whichever occurs first. Occurrence and date of disease progression in rwPFS will be determined from documentation within the patient record, such as pathology reports, imaging report notes, and statements about disease progression in the oncologist progress notes. Patients without an event (progression/death) will be censored at last date of assessment.
Overall survival | Retrospective: from date of first diagnosis of unresectable or mBC (01 January 2017) to the end of follow-up (i.e., until death, the last medical record entry, or date of data extraction, whichever is the earliest) [Approximately 12 Months]
  Length of time from the date of diagnosis of unresectable or mBC or date of initiation of LOT to death due to any cause. If patient is not dead until the last record available or date of data extraction, then time-to-event will be calculated for that date. Patients who are known to be alive at the date of data collection will be censored at the date of data collection. Patients who are lost to follow up will be censored on the date they were last known to be alive (eg. date of last recorded hospital visit).
Real-world objective response rate | Retrospective: from date of first diagnosis of unresectable or mBC (01 January 2017) to the end of follow-up (i.e., until death, the last medical record entry, or date of data extraction, whichever is the earliest) [Approximately 12 Months]
  The percentage of patients who have achieved real-world partial response (rwPR) and real-world complete response (rwCR) to therapy for each LOT.
Real-world disease control rate | Retrospective: from date of first diagnosis of unresectable or mBC (01 January 2017) to the end of follow-up (i.e., until death, the last medical record entry, or date of data extraction, whichever is the earliest) [Approximately 12 Months]
  The percentage of patients with rwCR, rwPR and real-world stable disease (rwSD) during treatment for each LOT
Percentage of Proportion of patients with AESIs that led to treatment discontinuations, hospitalisatons and deaths. | Retrospective: from date of first diagnosis of unresectable or mBC (01 January 2017) to the end of follow-up (i.e., until death, the last medical record entry, or date of data extraction, whichever is the earliest) [Approximately 12 Months]
  Assessment of safety and tolerability of different treatment regimens in patients with HER2-positive unresectable or mBC.

CONTACTS AND LOCATIONS:
Locations (32):
- Australia (5):
  - Research Site, Macquarie, New South Wales
  - Research Site, Newcastle, New South Wales
  - Research Site, Parramatta, New South Wales
  - Research Site, St Leonards, New South Wales
  - Research Site, Perth, Western Australia
- Brazil (13):
  - Research Site, Manaus, Amazonas
  - Research Site, Fortaleza, Ceará
  - Research Site, Cachoeiro de Itapemirim, Espírito Santo
  - Research Site, Salvador, Estado de Bahia
  - Research Site, Curitiba, Paraná
  - Research Site, Caxias do Sul, Rio Grande do Sul
  - Research Site, Porto Alegre, Rio Grande do Sul
  - Research Site, Itajaí, Santa Catarina
  - Research Site, Santo André, São Paulo
  - Research Site, Fortaleza
  - Research Site, Goiânia
  - Research Site, Rio de Janeiro
  - Research Site, São Paulo
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, Kowloon
- Singapore (3):
  - Research Site, Singapore, Central Singapore
  - Research Site, Singapore, South East
  - Research Site, Singapore
- South Korea (4):
  - Research Site, Incheon, Incheon Gwang Yeogsi
  - Research Site, Seoul, Seoul Teugbyeolsi
  - Research Site, Goyang
  - Research Site, Seoul
- Taiwan (5):
  - Research Site, Tainan County, Tainan
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com /ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com /ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at:
  https://astrazenecagrouptrials.pharmacm.com /ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9673R00005&attachmentIdentifier=4e22cdbe-b63e-49bf-b8fd-9d606ff71604&fileName=D9673R00005_PXL_253938_Draft_1_CSR_Synopsis_Redacted_04Jul24_For_AZCT.pdf&versionIdentifier=